CLINICAL TRIAL: NCT07337473
Title: Effect of Evidence-based Digital Cognitive Behavior Therapy for Adolescents With Nonsuicidal Self-Injury Disorder: A Randomized Clinical Trial
Brief Title: Evidence-based Digital CBT for Nonsuicidal Self-Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Sixth Hospital (Other)
Responsible Party: Principal Investigator, Yi Zhong, Peking University, Peking University Sixth Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PekingUSH 20251020
Record Dates: First submitted 2025-11-30; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Non Suicidal Self Injury; Cognitive Behavior Therapy
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based digital CBT group (Experimental): Participants will receive 6 weeks of evidence-based digital cognitive behaviour therapy, adjunctive to treatment as usual, as provided in the community or research group.
  Interventions: Behavioral: Evidence-based digital cognitive behaviour therapy
- Health Education group (Active Comparator): Participants will receive health education for 6 weeks, adjunctive to treatment as usual, as provided in the community or research group.
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Evidence-based digital cognitive behaviour therapy — The Evidence-based digital cognitive behaviour therapy is delivered via an internet platform during the intervention period via the platform.
  Arms: Evidence-based digital CBT group
Behavioral: Health Education — The Health Education therapy is delivered via an internet platform during the intervention period via the platform.
  Arms: Health Education group

SUMMARY:
To evaluate if evidence-based digital cognitive behaviour therapy for adolescents is an efficacious treatment when delivered as an adjunctive treatment to treatment as usual, compared to a control group consisting of treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* 5 nonsuicidal self-injury episodes past year
* 1 nonsuicidal self-injury episodes past month having at least one parent who committed to participate in the program

Exclusion Criteria:

Severe suicidal ideation a diagnosis of psychotic or ongoing (past month) substance dependence the presence of co-occurring psychological disorders that required immediate treatment (i.e., severe anorexia nervosa)

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Ottawa Self-injury Inventory（OSI） | From the date of baseline assessment (enrollment) until the date of 12-month follow-up, assessed at baseline, post-treatment (Day 1 of the week following treatment completion), and 1 month, 6 months, and 12 months after post-treatment.
  Assessing the frequency and severity of nonsuicidal self-injury

SECONDARY OUTCOMES:
General Anxiety Disorder-7 | Change from baseline (Day 1 of study enrollment), assessed every 2 weeks during the 6-week treatment period, at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  GAD-7 total score for the seven items ranges from 0 to 21. 0-4: minimal anxiety. 5-9: mild anxiety. 10-14: moderate anxiety. 15-21: severe anxiety.
Patient Health Questionnaire-9 | Change from baseline (Day 1 of study enrollment), assessed every 2 weeks during the 6-week treatment period, at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used brief screening tool that can assist both in identifying individuals with major depression disorder, as well as assessing the severity of depressive symptoms.
Beck's Suicide Intent Scale | Change from baseline (Day 1 of study enrollment), assessed every week during the 6-week treatment period, at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  The total score of the BSSI ranges from 0 to 37, with higher scores indicating more severe suicidal ideation
Self-harm behaviour craving visual analog scale | Change from baseline (Day 1 of study enrollment), assessed every week during the 6-week treatment period, at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  Assessment of self-harm behaviour craving in NSSI adolescent
Difficulties in Emotion Regulation Scale - 16-item version (DERS) | Change from baseline (Day 1 of study enrollment), assessed at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  Difficulties in emotion regulation. Higher scores indicate more difficulties.

OTHER OUTCOMES:
Internet Addiction Test | Change from baseline (Day 1 of study enrollment), assessed at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  The IAT total score is the sum of the ratings given by the examinee for the 20 item responses. Each item is rated on a 5-point scale ranging from 0 to 5. The maximum score is 100 points. The higher the score is, the higher is the severity of your problem. Total scores that range from 0 to 30 points are considered to reflect a normal level of Internet usage; scores of 31 to 49 indicate the presence of a mild level of Internet addiction; 50 to 79 reflect the presence of a moderate level; and scores of 80 to 100 indicate a severe dependence upon the Internet.
The Pittsburgh Sleep Quality Index | Change from baseline (Day 1 of study enrollment), assessed at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties
Insomnia Severity Index | Change from baseline (Day 1 of study enrollment), assessed every 2 weeks during the 6-week treatment period, at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  Respondents rate each element of the questionnaire using Likert-type scales. Responses can range from 0 to 4, where higher scores indicate more acute symptoms of insomnia. Scores are tallied and can be compared both to scores obtained at a different phase of treatment and to the scores of other individuals. Though developers point out that their chosen cutoff scores have not been validated, they offer a few guidelines for interpreting scale results: a total score of 0-7indicates"no clinically significant insomnia, "8-14 means"subthreshold insomnia, "15-21 is"clinical insomnia(moderate severity), "and 22-28 means"clinical insomnia(severe). "
The Morningness-Eveningness Questionnaire (MEQ)-5 | Change from baseline (Day 1 of study enrollment), assessed at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  Assess morningness and eveningness. Questions are framed in a preferential manner, where the respondent is asked to indicate when, for example, he/she would prefer to wake up or start sleep, rather than when he/she actually does.
Dysfunctional Beliefs and Attitudes about Sleep (DBAS) | Change from baseline (Day 1 of study enrollment), assessed at post-treatment (Day 1 of the week following treatment completion), and at 1 month, 6 months, and 12 months after post-treatment.
  The Dysfunctional Beliefs about Sleep Scale - short version (DBAS-16) is a self-report questionnaire designed to assess beliefs, attitudes, and misconceptions about sleep that may contribute to insomnia. It consists of 16 items that measure various cognitive distortions related to sleep, such as unrealistic expectations, misattributions about insomnia, and concerns about the consequences of poor sleep

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the research results, the data will be shared on this website and relevant journal platforms
Supporting Information: Study Protocol

REFERENCES:
- [Result] Bjureberg J, Ojala O, Hesser H, Habel H, Sahlin H, Gratz KL, Tull MT, Claesdotter Knutsson E, Hedman-Lagerlof E, Ljotsson B, Hellner C. Effect of Internet-Delivered Emotion Regulation Individual Therapy for Adolescents With Nonsuicidal Self-Injury Disorder: A Randomized Clinical Trial. JAMA Netw Open. 2023 Jul 3;6(7):e2322069. doi: 10.1001/jamanetworkopen.2023.22069. PMID 37440232
- [Result] Morthorst B, Olsen MH, Jakobsen JC, Lindschou J, Gluud C, Heinrichsen M, Mohl B, Rubaek L, Ojala O, Hellner C, Bjureberg J, Pagsberg AK. Internet based intervention (Emotion Regulation Individual Therapy for Adolescents) as add-on to treatment as usual versus treatment as usual for non-suicidal self-injury in adolescent outpatients: The TEENS randomised feasibility trial. JCPP Adv. 2022 Dec 3;2(4):e12115. doi: 10.1002/jcv2.12115. eCollection 2022 Dec. PMID 37431416
- [Result] Kaess M, Edinger A, Fischer-Waldschmidt G, Parzer P, Brunner R, Resch F. Effectiveness of a brief psychotherapeutic intervention compared with treatment as usual for adolescent nonsuicidal self-injury: a single-centre, randomised controlled trial. Eur Child Adolesc Psychiatry. 2020 Jun;29(6):881-891. doi: 10.1007/s00787-019-01399-1. Epub 2019 Sep 11. PMID 31512050
- [Result] Franklin JC, Fox KR, Franklin CR, Kleiman EM, Ribeiro JD, Jaroszewski AC, Hooley JM, Nock MK. A brief mobile app reduces nonsuicidal and suicidal self-injury: Evidence from three randomized controlled trials. J Consult Clin Psychol. 2016 Jun;84(6):544-57. doi: 10.1037/ccp0000093. Epub 2016 Mar 28. PMID 27018530